CLINICAL TRIAL: NCT00801060
Title: A Phase 2, Randomized, Open-Label Study to Evaluate the Safety and Efficacy of Fludarabine, Cyclophosphamide, and Rituximab (FCR) in Combination With Lumiliximab Versus FCR Alone in Subjects With Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Evaluation of Safety and Efficacy of Fludarabine, Cyclophosphamide, and Rituximab (FCR) +/- Lumiliximab in Subjects With Previously Untreated Chronic Lymphocytic Leukemia (CLL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 152CL202; EUDRACT NO: 2008-002204-25
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Fludara; CD23; Cyclophosphamide; Antibody; Fludarabine; CLL; Rituximab; Mabthera; Biogen Idec; Lumiliximab; Rituxan; Cytoxan; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — lumiliximab; Receptors, Fc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group A (Experimental): FCR + Lumiliximab (L)
  L (Lumiliximab): Day 2 50 mg/m2, Day 4 450 mg/m2, for the first week, then single doses of 500 mg/m2 every four weeks, for 21 weeks.
  F (Fludarabine): 25 mg/m2 daily, every four weeks for 21 weeks
  C (Cyclophosphamide): 250 mg/m2 daily, every four weeks for 21 weeks
  R: (Rituximab): Day 1 50 mg/m2, Day 3 325 mg/m2, for the first week, then single doses of 500 mg/m2 every four weeks, for 21 weeks
  Interventions: Drug: Lumiliximab + FCR
- Treatment Group B (Active Comparator): FCR
  F (Fludarabine): 25 mg/m2 daily, every four weeks for 21 weeks
  C (Cyclophosphamide): 250 mg/m2 daily, every four weeks for 21 weeks
  R: (Rituximab): Day 1 50 mg/m2, Day 3 325 mg/m2, for the first week, then single doses of 500 mg/m2 every four weeks, for 21 weeks
  Interventions: Drug: FCR

INTERVENTIONS:
Drug: Lumiliximab + FCR — Dose, schedule, and duration in the protocol
  Arms: Treatment Group A
Drug: FCR — Dosage, schedule, and duration in the protocol
  Arms: Treatment Group B

SUMMARY:
This is a Phase 2, randomized, open-label, multicenter study in subjects with previously untreated CLL. It is designed to evaluate safety and efficacy of fludarabine, cyclophosphamide, rituximab (FCR) and lumiliximab versus FCR alone.

DETAILED DESCRIPTION:
See protocol.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 18 years or older.
* Previously untreated CD23+ and CD20+ B cell CLL.
* Life expectancy >6 months.
* Subjects with Rai Stage III or IV (Binet Stage C) or Rai Stage I or II (Binet Stage A or B) if determined to have active disease.
* World Health Organization (WHO) Performance Status ≤2.
* Normal ECG with QTc ≤450 msec for men and ≤460 msec for women. PR interval (Print) must be <240 msec and QRS complex <110 msec. T wave flattening and T wave inversion will be permitted.
* All male subjects and female subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 12 months after their last dose of study treatment.
* Acceptable liver function at Screening.
* Acceptable hematologic status at Screening.
* Acceptable renal function at Screening.
* Subjects receiving any medication known to affect the QTc interval must discontinue the use of the medication or be on a stable dose of the medication for at least 3 months or 5 half-lives (whichever is longer) prior to Study Day 1, and continue (whenever possible) at the same dose throughout the study.

EXCLUSION CRITERIA:

* Any prior therapy for CLL.
* Known history or positive test result for human immunodeficiency virus.
* Known history of, or positive test result for Hepatitis C virus (test for Hepatitis C virus antibody) or Hepatitis B virus (test for Hepatitis B Surface Antigen and Hepatitis B Core Antibody) at Screening.
* Uncontrolled diabetes mellitus.
* Uncontrolled hypertension.
* Hypokalemia.
* Hypomagnesemia.
* New York Heart Association Class III or IV cardiac disease; myocardial infarction within the past 6 months prior to Study Day 1.
* Arrhythmia (other than sinus arrhythmia) within 30 days prior to Study Day 1.
* Evidence of active myocardial ischemia on ECG.
* Subjects with pacemakers.
* Transformation to aggressive B-cell malignancy.
* Secondary malignancy requiring active treatment.
* Any medical condition that would require long-term use (>1 month) of systemic corticosteroids during study treatment.
* Any serious nonmalignant disease or laboratory abnormality, which would confound the evaluation of adverse events (AEs).
* Active bacterial, viral, or fungal infections.
* Any known family history of long QT syndrome.
* Seizure disorders requiring anticonvulsant therapy.
* Severe chronic obstructive pulmonary disease with hypoxemia.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Study Day 1.
* Clinically active autoimmune disease.
* Presence of history of Coombs positive hemolytic anemia.
* Pregnant or currently breastfeeding at Screening.
* Prior exposure to lumiliximab or any other anti CD23 antibody.
* Subjects with known hypersensitivity to Chinese hamster ovary cell proteins, murine proteins, or any component of fludarabine, cyclophosphamide, rituximab, or the lumiliximab investigational treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of FCR+L compared with FCR alone in subjects with previously untreated CLL. | June 2010
To evaluate the efficacy of FCR+L compared with FCR alone in subjects with previously untreated CLL. | June 2010

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (34):
- United States (9):
  - University of Florida/Pulmonary, Critical Care & Sleep Medicine, Gainesville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Research Site, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Research Site, Detroit, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Research Site, Hackensack, New Jersey
  - Vanderbilt University Medical Center-IPF Program, Nashville, Tennessee
  - Research Site, Seattle, Washington
- Australia (2):
  - Research Site, Westmead, New South Wales
  - Research Site, Melbourne (Coburg), Victoria
- Austria (2):
  - Research Site, Graz
  - Research Site, Vienna
- Belgium (6):
  - Research Site, Antwerp
  - Research Site, Brussels
  - Research Site, Leuven
  - Research Site, Mont-Godinne
  - Research Site, Roeselare
  - Research Site, Wilrijk
- Research Site, Ottawa, Ontario, Canada
- France (7):
  - Research Site, Paris, Cedex
  - Research Site, Pierre-Bénite, Cedex
  - Research Site, Lille
  - Research Site, Montpellier
  - Research Site, Pessac
  - Research Site, Strasbourg
  - Research Site, Tours
- Poland (3):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Lodz
- United Kingdom (4):
  - Research Site, Exeter, Devon
  - Research Site, Plymouth, Devon
  - Research Site, London, England
  - Research Site, Bath, Avon